CLINICAL TRIAL: NCT03337321
Title: Developing and Validating Digital Affective Patient Experience/Outcome Measure
Acronym: ETVa
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Aalto University (Other)
Responsible Party: Principal Investigator, Maritta Poyhonen-Alho, Principal Investigator, Helsinki University Central Hospital
Other Study IDs: 2329/2016
Record Dates: First submitted 2017-10-17; First posted 2017-11-09 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Affective; Reaction; Pregnancy Related; Validation Studies
Keywords: pregnancy; emotions; patient experience; maternal care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ETvalid: Pregnant women attending maternal care services and having access to computational device

SUMMARY:
The aim of the research project is to develop and validate a new digital measure of affective patient experience in maternal care. In this validating study extensive collection of affective ratings of 195 emotion words is collected. Pregnant women at different gestational stages are asked to provide affective ratings of 195 emotion words in relation to the dimensions: pleasure, arousal, dominance. Based on these ratings population averages and properties of emotion words will be calculated. The measure will be developed in respect to the analysis of affective rating and supplementing data.

DETAILED DESCRIPTION:
As there is an increasing demand for and interest in measures that take patient's emotions into account, this research project aims to develop and validate a new digital measure of affective patient-reported experience/outcome in maternal care.

In this validating study extensive collection of affective ratings of 195 emotion words will be collected. Pregnant women (N=1000) at different gestational stages are asked to provide affective ratings of 195 emotion words in relation to the dimensions: pleasure, arousal, dominance. This is done by using a visual Likert scale (Self-Assessment Manikin). The pregnant women participating in the research are also asked to answer to various questionnaires to identify patterns of personality, behavior and the state of health and well-being. Based on the affective ratings population averages and properties of emotion words will be calculated. The measure will be developed in respect to the analysis of affective ratings and supplementing data.

The research provides insights on how affective ratings could be connected to clinical indicators and patient experience.

ELIGIBILITY:
Inclusion Criteria:

* ongoing pregnancy
* attending maternal care in the Hospital District of Helsinki and Uusimaa
* fluent in Finnish
* access to mobile communication device

Exclusion Criteria: none

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: Pregnant women attending maternal care in the Hospital District of Helsinki and Uusimaa
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-13 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
three-dimensional affective ratings | 9 months
  affective rating of 195 emotion words in relation to pleasure, arousal, dominance (Lang 1980)

SECONDARY OUTCOMES:
anxiety | 9 months
  Generalized Anxiety Disorder Scale (GAD-7) (Spitzer et al. 2006). Scale is from 0 to 21. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.

OTHER OUTCOMES:
S5 personality traits (30 facets of the Five-Factor Model) | 9 months
  Short Five S5, a 60-item questionnaire (Konstabel et al 2012), is used to measure personality traits, more specifically, the 30 facets of the Five-Factor Model, using comprehensive single items (CSI).
emotion regulation | 9 months
  State and Trait meta-mood questionnaire (adapted from: Mayer & Stevens 1994; Salovey et al 1995)
health related quality of life | 9 months
  PROMIS-10 (Cella et al 2007)
emotional stress reaction | 9 months
  Emotional Stress Reaction Questionnaire (ESRQ) (Larsson&Wilde-Larsson 2010)
subjective well-being | 9 months
  Subjective Well-Being Questionnaire (SWB) (Lee et al 2013)
patient experience in maternal care | 9 months
  Pregnancy- and maternity-care patients' experiences questionnaire (PreMaPeq) (Sjetne et al 2015)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital District of Helsinki and Uusimaa, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lang, P. J. (1980). Behavioral treatment and bio-behavioral assessment: computer applications. In J. B. Sidowski, J. H. Johnson, & T. A. Williams (Eds.), Technology in mental health care delivery systems (pp. 119-l37). Norwood, NJ: Ablex.
- [Background] Konstabel, K., Lönnqvist, J.-E., Walkowitz, G., Konstabel, K. and Verkasalo, M. (2012), The 'Short Five' (S5): Measuring personality traits using comprehensive single items. European Journal of Personality, 26(1), 13-29. doi:10.1002/per.813
- [Background] Mayer, J., & Stevens, A. (1994). An emerging understanding of the reflective (meta-) experience of mood. Journal of Research in Personality, 28, 351-373.
- [Background] Salovey, P., Mayer, J. D., Goldman, S. L., Turvey, C., and Palfai, T. P. (1995). Emotional attention, clarity, and repair: Exploring emotional intelligence using the Trait Meta-Mood Scale. In J. W. Pennebaker (Ed.), Emotion, Disclosure and Health (pp.125-151). Washington, DC: American Psychological Association.
- [Background] Cella D, Yount S, Rothrock N, Gershon R, Cook K, Reeve B, Ader D, Fries JF, Bruce B, Rose M; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS): progress of an NIH Roadmap cooperative group during its first two years. Med Care. 2007 May;45(5 Suppl 1):S3-S11. doi: 10.1097/01.mlr.0000258615.42478.55. PMID 17443116
- [Background] Larsson G, Wilde-Larsson B. Quality of care and patient satisfaction: a new theoretical and methodological approach. Int J Health Care Qual Assur. 2010;23(2):228-47. doi: 10.1108/09526861011017120. PMID 21388102
- [Background] Lee H, Vlaev I, King D, Mayer E, Darzi A, Dolan P. Subjective well-being and the measurement of quality in healthcare. Soc Sci Med. 2013 Dec;99:27-34. doi: 10.1016/j.socscimed.2013.09.027. Epub 2013 Oct 8. PMID 24355467
- [Background] Sjetne IS, Iversen HH, Kjollesdal JG. A questionnaire to measure women's experiences with pregnancy, birth and postnatal care: instrument development and assessment following a national survey in Norway. BMC Pregnancy Childbirth. 2015 Aug 21;15:182. doi: 10.1186/s12884-015-0611-3. PMID 26294064
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- See also: The Institute of Healthcare Engineering, Management and Architecture (the HEMA Institute) at Aalto University School of Science, Finland — http://hema.aalto.fi/en/